CLINICAL TRIAL: NCT02644395
Title: Thiazide Diuretics for Hypertension in Kidney Transplant Recipients Using Tacrolimus
Acronym: TT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Associate Professor, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2012-417
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Hypertension; Kidney Transplantation
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine (Active Comparator): Current treatment of choice
  Interventions: Drug: Amlodipine
- Chlorthalidone (Experimental): Testing new indication for approved drug
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Chlorthalidone — Drug
  Arms: Chlorthalidone
Drug: Amlodipine — Drug
  Arms: Amlodipine

SUMMARY:
Background: Calcineurin inhibitors (CNIs) are the most commonly used immunosuppressive drugs to prevent rejection after kidney transplantation. However, the efficacy of preventing rejection comes at the cost of important side-effects. Among the most common side-effects is hypertension. Hypertension after kidney transplantation is clinically relevant, because it increases the risk of cardiovascular disease and is associated with increased graft loss and recipient mortality. The mechanism of CNI-induced hypertension is incompletely understood and, therefore, the treatment is currently empiric. These and other investigators recently showed that CNIs cause salt-sensitive hypertension by activating a sodium transporter in the kidney, namely the thiazide-sensitive sodium chloride cotransporter.

Hypothesis: The investigators hypothesize that thiazide diuretics are non-inferior to calcium channel blockers (CCBs) (currently usually the treatment of choice) for the treatment of CNI-induced hypertension.

Objective: To compare the blood pressure response to thiazide diuretics and CCBs in patients with CNI-induced hypertension.

Study design: Single-center, randomized cross-over trial.

Study population: Kidney transplant recipients with a good functioning allograft (eGFR > 30 ml/min) who are hypertensive (daytime systolic blood pressure > 140 mm Hg) and who do not have proteinuria (< 1 g/day).

Intervention: Patients will be randomized to receive chlorthalidone (12.5 mg once daily, if needed titrated to 25 mg once daily) or amlodipine (5 mg once daily, if needed titrated to 10 mg once daily).

Main study parameters/endpoints: 24-hour blood pressure recording.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both drugs have long been registered for the treatment of hypertension. The side-effect profile of both drugs is considered to be equal. The burden of the study for the patients are blood pressure measurements using 30-minute automated blood pressure measurement and 24-hour ambulatory blood pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients using tacrolimus
* Average daytime SBP > 140 mm Hg (ABPM)
* eGFR > 30 ml/min (MDRD)

Exclusion Criteria:

* Use of glucocorticoids, co-trimoxazole, diuretics
* Pregnancy
* Serum sodium < 136, serum potassium < 3.5
* Proteinuria > 1 g/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Average daytime SBP | 8 weeks

SECONDARY OUTCOMES:
Laboratory parameters | 8 weeks
Side effects | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, Netherlands

REFERENCES:
- [Background] Moes AD, Hesselink DA, van den Meiracker AH, Zietse R, Hoorn EJ. Chlorthalidone Versus Amlodipine for Hypertension in Kidney Transplant Recipients Treated With Tacrolimus: A Randomized Crossover Trial. Am J Kidney Dis. 2017 Jun;69(6):796-804. doi: 10.1053/j.ajkd.2016.12.017. Epub 2017 Mar 1. PMID 28259499
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471